CLINICAL TRIAL: NCT02941094
Title: Insertion Angle and Needle Visualization During Ultrasound Guided Internal Jugular Vein Cannulation
Acronym: US_angle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: refa-US-angle
Record Dates: First submitted 2016-07-19; First posted 2016-10-21 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Internal Jugular Vein Cannulation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- angle 30 group (Active Comparator): During central line insertion, After choosing the proper position, the skin was infiltrated with %1 lidocaine. The vein will be localized using linear ultrasound probe (PLT-805AT, 8 MHz, Toshiba Tokyo, Japan) attached to ultrasound machine (Xario, Toshiba Tokyo Japan). The needle will be advanced guided by the ultrasound probe with needle skin angle 30-40 degree.
  Interventions: Device: needle PLT-805AT; Device: Ultrasound
- angle 50 group (Active Comparator): During central line insertion,After choosing the proper position, the skin was infiltrated with %1 lidocaine. The vein will be localized using linear ultrasound probe (PLT-805AT, 8 MHz, Toshiba Tokyo, Japan) attached to ultrasound machine (Xario, Toshiba Tokyo Japan). The needle will be advanced guided by the ultrasound probe with needle skin angle 50-60 degree
  Interventions: Device: needle PLT-805AT; Device: Ultrasound
- angle 70 group (Active Comparator): During central line insertion,After choosing the proper position, the skin was infiltrated with %1 lidocaine. The vein will be localized using linear ultrasound probe (PLT-805AT, 8 MHz, Toshiba Tokyo, Japan) attached to ultrasound machine (Xario, Toshiba Tokyo Japan). The needle will be advanced guided by the ultrasound probe with needle skin angle 60-80 degree
  Interventions: Device: needle PLT-805AT; Device: Ultrasound

INTERVENTIONS:
Device: needle PLT-805AT — comparing success rate and complications using different needle to US probe angles.
  Other Names: PLT-805AT, 8 MHz, Toshiba Tokyo, Japan
Device: Ultrasound — Xario, Toshiba Tokyo Japan

SUMMARY:
Ultrasound guidance has been established as an effective and safe method during insertion of internal jugular vein catheter.. Needle visualization during advancement toward the vein has a great impact on both safety and success of the procedure. Clinicians have adopted variable techniques to increase needle visualization including changing needle- probe relation (in-plane vs. out-of-plane), or using specific ultrasound needles The angle between the inserting needle and the probe lying on patient skin affects both the distance to the vein and the length of the needle part travelling through the us beam

ELIGIBILITY:
Inclusion Criteria:

* all patients requiring central line insertion

Exclusion Criteria:

* refusal
* coagulopathy
* neck surgeries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
success rate | 24 hours starting from central line insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided